CLINICAL TRIAL: NCT03799653
Title: A Prospective Cohort Study of Common Chronic Diseases on Nurses in Xiamen, China: Nurse Cohort Study Xiamen (NCSX)
Brief Title: A Nurse Cohort Study in Xiamen, China
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Zhibin LI, Director, The First Affiliated Hospital of Xiamen University
Other Study IDs: KYH2019-002
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma and urin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses: All subjects are registered nurses in Xiamen, China
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a prospective observational study, and there is no intervention.

SUMMARY:
The Nurse Cohort Study Xiamen (NCSX) is an open-ended prospective cohort study with very broad research aims. The primary objectives of the NCSX is planned to examine genetic, epigenetic, biological, psychological, social, lifestyle and other environmental factors of nurses in relation to incidence and progression of the common chronic diseases, such as hypertension, ischemic heart disease, stroke, diabetes, chronic kidney disease and some cancers, which are emerging with economic development in Xiamen, China. Specifically, we intend to test whether empirically driven hypothesis and emerging risk factors mainly developed in response to observations in economically developed Western societies apply in a population living in a rapid changing lifestyle in China now.

DETAILED DESCRIPTION:
Objectives: To establish a cohort of about 10,000 registered nurses (aged 20 or over) in Xiamen, China; to describe the baseline major risk factors; to analyze their interrelationships; and to examine the risks of incidence and progression of major chronic diseases, such as hypertension, stroke, CKD and cancers, and all-cause and cause-specific mortality by different levels of the risk factors after about 5 years follow-up.

Design: A prospective cohort study. Setting: 7 public hospitals in Xiamen, China. Participants: About 10,000 registered nurses (aged 20 or over) who work in public hospitals in Xiamen, China.

Main outcome: Incidences of common chronic diseases, such as CVD, diabetes, chronic kidney disease, and cancers; progression of these diseases; all cause and specific-cause mortality.

Hypothesis: Relative risks of major risk factors. Results of the study should have strong impact on prevention and control of these diseases and promoting nurses'health in the local population.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses of public hospitals in Xiamen, China;
* aged 20 years or over;
* Working in the public hospitals for at least 1 year;
* Signed the informed consent and agreed to participate in the study;
* Assuming not moved out of Xiamen for at least 5 years;

Exclusion Criteria:

* who are unambulatory;
* who are receiving treatment modalities, which , if omitted, may result in immediate life threatening risk such as chemotherapy or radiotherapy for cancer, or dialysis for renal failure.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Registered nurses in public hospitals in Xiamen, China;
  * Aged 20 years or over and living in Xiamen for at least 1 year and will not move out of Xiamen for at least 5 years;
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate | 2019.1.21-2024.12.31
  The incidence rates of common chronic diseases, such as hypertension, The stroke, CKD and cancers

SECONDARY OUTCOMES:
Mortality | 2019.1.21-2024.12.31
  All-cause and cause-specific mortality

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Li, Ph.D., Study Chair — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided